CLINICAL TRIAL: NCT03111147
Title: The Impact of Humeral Component Version on Outcomes Following Reverse Total Shoulder Arthroplasty: A Prospective Randomized Controlled Trial
Brief Title: Impact of Humeral Component Version on Outcomes Following RTSA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Michael Wiater, ◾Vice Chairman Orthopedic Surgery◾Chief of Shoulder Surgery ◾Program Director, Fellowship in Shoulder and Elbow Surgery ◾Program Director, Orthopaedic Surgery Residency, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-057
Record Dates: First submitted 2017-04-07; First posted 2017-04-12 (Actual); Results first posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Rotator Cuff Tear Arthropathy
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 0 degrees humeral component version (Experimental): Reverse Total Shoulder Arthroplasty with humeral component positioned in 0 degrees of version
  Interventions: Device: 0 degrees humeral component version
- 30 degrees humeral component retroversion (Experimental): Reverse Total Shoulder Arthroplasty with humeral component positioned in 30 degrees of retroversion
  Interventions: Device: 30 degrees humeral component retroversion

INTERVENTIONS:
Device: 0 degrees humeral component version — RTSA with humeral component positioned in 0 degrees of version
  Arms: 0 degrees humeral component version
Device: 30 degrees humeral component retroversion — RTSA with humeral component positioned in 30 degrees of retroversion
  Arms: 30 degrees humeral component retroversion

SUMMARY:
The proposed study is a prospective, single-blinded, randomized trial to investigate the impact of humeral component version on shoulder range of motion and patient reported functional outcomes following reverse total shoulder arthroplasty.

DETAILED DESCRIPTION:
Retrospective clinical evidence suggests that increasing humeral component retroversion does not affect measured internal or external rotation, however patients with neutral version may experience better function with daily activities requiring internal rotation compared to those with 30 degrees of retroversion. Prospective data on clinical outcomes comparing different humeral component versions in RTSA is currently lacking. The proposed study is a prospective, single-blinded, randomized trial to investigate the impact of humeral component version on shoulder range of motion and patient reported functional outcomes following reverse total shoulder arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary reverse total shoulder arthroplasty
* Diagnosis of cuff tear arthropathy or primary OA with RCT
* Intact posterior rotator cuff and subscapularis preoperatively, as determined by surgeon-administered physical exam
* 18 years or older

Exclusion Criteria:

* Revision arthroplasty
* Diagnosis of rheumatoid arthritis, infection, acute trauma or instability
* Minors (under 18 years of age)

  * Prior open shoulder surgery
  * Concomitant latissimus dorsi transfer
  * Patients not undergoing a standard of care physical therapy protocol
  * Pregnant, patient-reported
  * Cognitively impaired

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2023-05-23 (Actual); Study Completion 2023-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Michael Wiater, MD, Principal Investigator — Corewell Health East
Locations (1):
- Beaumont Health, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 95 patients recruited, 85 met inclusion criteria and were randomized to treatment groups.
Period: Overall Study
Arm/Group | 0 Degrees Humeral Component Version | 30 Degrees Humeral Component Retroversion
Started | 42 | 43
Completed | 33 | 33
Not Completed | 9 | 10
Not completed — Lost to Follow-up | 2 | 5
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Protocol Violation | 2 | 1
Not completed — Death | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0 Degrees Humeral Component Version | 30 Degrees Humeral Component Retroversion | Total
Number analyzed (Participants) | 42 | 43 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.20 (8.21) | 69.19 (7.45) | 69.19 (7.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 31 | 54
  Male | 19 | 12 | 31
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 42 | 43 | 85

OUTCOME MEASURES:

1. Primary Outcome: Postoperative External Range of Motion (ROM)
Description: External range of motion measurements of the shoulder in degrees
Time Frame: 2 years
Population: 9 participants in the 0 degrees humeral component version and 10 patients in the 30 degrees humeral component retroversion did not complete study activities and no data was collected.
Measure: Mean (Standard Error); unit: degrees
Arm/Group | 0 Degrees Humeral Component Version | 30 Degrees Humeral Component Retroversion
Number analyzed (Participants) | 33 | 33
degrees | 35 (3.4) | 39 (2.1)

2. Primary Outcome: Postoperative Internal Range of Motion (ROM)
Description: Internal range of motion measurements of the shoulder in degrees
Time Frame: 2 years
Population: as for outcome 1
Measure: Mean (Standard Error); unit: degrees
Arm/Group | 0 Degrees Humeral Component Version | 30 Degrees Humeral Component Retroversion
Number analyzed (Participants) | 33 | 33
degrees | 35.5 (3.2) | 33.5 (2.5)

ADVERSE EVENTS:
Time Frame: 2 years
Description: Only shoulder related adverse events were assessed and collected per protocol
Arm/Group | 0 Degrees Humeral Component Version | 30 Degrees Humeral Component Retroversion
All-Cause Mortality (participants affected / at risk) | 1/42 | 1/43
Serious Adverse Events (participants affected / at risk) | 1/42 | 3/43
Other Adverse Events (participants affected / at risk) | 11/42 | 9/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0 Degrees Humeral Component Version (N=42) | 30 Degrees Humeral Component Retroversion (N=43)
Revision Reverse Total Shoulder Arthroplasty (Surgical and medical procedures) | 0 (0) | 2 (2)
COVID Infection resulting in Death (Infections and infestations) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0 Degrees Humeral Component Version (N=42) | 30 Degrees Humeral Component Retroversion (N=43)
Heteroptopic ossification on inferior glenoid (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 7 (7)
Impingement (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Crepitus (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Inferior Scapular Notching (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Interval Bony Healing (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chronic changes to the distal acronium (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
New onset shoulder weakness (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Scapular spine tenderness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tendinitis (Deltoid) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Fracture (Scapular body) (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Numbness (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Brachioplexopathy (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Limited Range of Motion (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Muscle Spams (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
shoulder injury (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
humeral head subluxed inferiorly (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
elevated C-reactive protein (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
shoulder aspiration (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lateral deltoid insertion pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Shoulder strain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lucency around stem of humeral component (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
ecchymosis of proximal arm (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
new onset instability (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
positive sulcus sign (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
cortisone injection (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-02-08): https://cdn.clinicaltrials.gov/large-docs/47/NCT03111147/Prot_SAP_000.pdf
  • Informed Consent Form (2022-02-16): https://cdn.clinicaltrials.gov/large-docs/47/NCT03111147/ICF_001.pdf